CLINICAL TRIAL: NCT06138067
Title: A Pilot Study of Low Versus High Intensity Patient Navigation Program to Improve the Enrollment on Clinical Trials Among Cancer Patients
Brief Title: Patient Navigation Program to Improve Clinical Trial Enrollment in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: WellSpan Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: J23132; IRB00412107 (Other: JHM IRB)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Kidney Cancer
Keywords: clinical trials enrollment rate
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Approach (Experimental): Patients will receive printed educational material (PEM) which will include information and resources regarding clinical trials/clinical trial participation, cancer center support services; and community resources and services available to cancer patients. The PEM will be reviewed by the clinical trial patient navigator with the patient prior to the clinic visit with the medical oncologist. If the patient is offered participation in a therapeutic clinical trial, the high intensity patient navigation begins. The patient navigator will arrange to meet with the patient to complete a needs assessment to identify and address barriers to trial participation within one week of the visit with the medical oncologist (and clinical trial offer).
  Interventions: Behavioral: High intensity approach
- Low Intensity Approach (Active Comparator): Patients will receive printed educational material (PEM) which will include information and resources regarding clinical trials/clinical trial participation and community resources and services available to cancer patients. The PEM will be reviewed by the patient navigator with the patient prior to the clinic visit with the medical oncologist.
  Interventions: Behavioral: Low intensity approach

INTERVENTIONS:
Behavioral: High intensity approach — PEM, cancer center support services material, and community resources and services available to cancer patients material. The PEM will be reviewed with the patient navigator before the participants appointment with the medical oncologist. If enrolled in a clinical trial, the patient navigator will call the participant biweekly, or more often if they are working to resolve any needs identified in the needs assessment) until the participant is successfully enrolled in the therapeutic clinical trial. The patient navigator will call the participant once weekly for 4 weeks, or less than 4 weeks in other cases including withdrawal from the clinical trial or this navigation study, disease progression, or death. The participant will receive a call 3 months after enrollment on the therapeutic clinical trial to complete the Exit Questionnaire
  Arms: High Intensity Approach
Behavioral: Low intensity approach — The participant will receive PEM, and community resources and services available to cancer patients material. The PEM will be reviewed with the patient navigator before the appointment with the medical oncologist. The patient navigator will call the participant 4 weeks after enrollment on the trial. The participant will receive a call 3 months after enrollment on the therapeutic clinical trial to complete the Exit Questionnaire
  Arms: Low Intensity Approach

SUMMARY:
The goal of this clinical trial is to test the utility of patient navigation by comparing high intensity patient navigation to low intensity navigation approaches to improving cancer trial enrollment of patients treated in academic and community cancer centers. Patient navigation is a strategy for increasing patients access to cancer care by helping the participant overcome barriers in the participants communities and within the health care system by providing a bridge between the patient and the health care system. The primary objective of this study is to determine if a high intensity patient navigation program will improve patients enrollment on clinical trial in comparison to a low intensity patient navigation. Participants who agree to participate and are eligible will be randomly assigned to either the high intensity or low intensity approach.

DETAILED DESCRIPTION:
This study is a pilot randomized two arm prospective study of a high versus low intensity patient navigation program with the primary endpoint of clinical trials enrollment rate between the 2 arms. The hypothesis of the study is that a high intensity patient navigation program will improve the enrollment rates on clinical trials. Candidates for this study will already have been identified by the patient navigator as being potentially eligible for a clinical trial. Randomization will be stratified by the type of site: community versus academic. There will be a single futility analysis after approximately 50% of the patients have been randomized and offered a clinical trial. Randomization and data capture will be via REDCap.

The primary endpoint of the study is the enrollment rate on clinical trials. With a sample size of 90 and conservatively assuming a clinical trial enrollment among clinical trial eligible patients of 50%, simulations show the investigators would be able to detect a 25% minimum difference (alternative 75% enrollment) in enrollment rates between the two groups with 84% power using a Z test of proportions with a one-sided alpha level of 0.10.

ELIGIBILITY:
1. Age ≥ 18 years
2. Patient with a current diagnosis of a primary solid tumor including: prostate cancer and kidney cancer
3. Being seen at the Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins University (JHU) or Wellspan Health Center
4. Available therapeutic trial for the patient as determined through pre-screening/medical record review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients from high intensity navigation program that enroll in clinical trials | 18 months
  Number of patients from high intensity patient navigation program that enroll in clinical trials versus the number of patients from low intensity patient navigation program that enroll in clinical trials.

SECONDARY OUTCOMES:
Acceptance rate | 12 months
  Acceptance rate of patients on the navigation study.
Retention rate | 18 months
  Retention rate of patients on the navigation study

OTHER OUTCOMES:
Number of different types of barriers to enrollment | 18 months
  To identify type of potential barriers and total quantity of each type to enrollment on clinical trial reported by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ged, MBBS, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Wellspan, Chambersburg, Pennsylvania